CLINICAL TRIAL: NCT02311686
Title: Identifying the Profile of the Main Non-oxidative Biomarkers of Alcohol (Ethyl Glucuronide, Ethyl Sulphate, Fatty Acid Ethyl Esters) After the Experimental Exposure to Increasing Doses of Alcohol in Adults.
Brief Title: Non-oxidative Metabolite Profiles After Increasing Doses of Ethanol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Clara Pérez, PhD, Parc de Salut Mar
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: Biomarcadores/PNSD/1
Record Dates: First submitted 2014-12-03; First posted 2014-12-08 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Alcohol Consumption; Healthy
Keywords: Ethanol; Fatty acid ethyl esters; Ethyl glucoronide; Ethyl sulphate; Pharmacokinetics
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 10 g ethanol (Experimental): Subjects will be required to drink a dilution of 31 mL of vodka in 369 mL of lemon-flavored water in 15 minutes.
  Interventions: Dietary Supplement: 10 g ethanol
- 20 g ethanol (Experimental): Subjects will be required to drink a dilution of 63 mL of vodka in 337 mL of lemon-flavored water in 15 minutes.
  Interventions: Dietary Supplement: 20 g ethanol
- 40 g ethanol (Experimental): Subjects will be required to drink a dilution of 125 mL of vodka in 275 mL of lemon-flavored water in 15 minutes.
  Interventions: Dietary Supplement: 40 g ethanol
- 60 g ethanol (Experimental): Subjects will be required to drink a dilution of 188 mL of vodka in 212 mL of lemon-flavored water in 15 minutes.
  Interventions: Dietary Supplement: 60 g ethanol
- 80 g ethanol (Experimental): Subjects will be required to drink a dilution of 250 mL of vodka in 150 mL of lemon-flavored water in 15 minutes.
  Interventions: Dietary Supplement: 80 g ethanol

INTERVENTIONS:
Dietary Supplement: 10 g ethanol — Alcohol single oral dose
  Other Names: Vodka Absolut®
  Arms: 10 g ethanol
Dietary Supplement: 20 g ethanol — Alcohol single oral dose
  Other Names: Vodka Absolut®
  Arms: 20 g ethanol
Dietary Supplement: 40 g ethanol — Alcohol single oral dose
  Other Names: Vodka Absolut®
  Arms: 40 g ethanol
Dietary Supplement: 60 g ethanol — Alcohol single oral dose
  Other Names: Vodka Absolut®
  Arms: 60 g ethanol
Dietary Supplement: 80 g ethanol — Alcohol single oral dose
  Other Names: Vodka Absolut®
  Arms: 80 g ethanol

SUMMARY:
The aim of the study is to study the profile of ethanol and non-oxidative biomarkers (ethyl glucuronide, ethyl sulphate and fatty acid ethyl esters) after experimental administration of increasing doses of alcohol in adult subjects.

DETAILED DESCRIPTION:
The abuse of alcohol causes serious health and social problems. Alcohol consumption can be monitored by detecting biomarkers. In current practice indirect biomarkers (mean corpuscular volume, transaminases, gammaglutamyl or carbohydrate-deficient transferrin) are used, although direct biomarkers of alcohol, including alcohol itself and metabolites also exist.

Biomarkers of alcohol consumption are used as tools to prevent health and social problems related with alcohol, allowing the identification of subjects at risk of abuse, dependence or withdrawal and to assess the efficacy of treatments for alcohol dependence.

Non-oxidative metabolites (ethyl glucuronide, ethyl sulphate and fatty acid ethyl esters) have longer biological half-life than ethanol and accumulate in tissues after consumption.

The objective of the study is to study the profile of ethanol and non-oxidative biomarkers (ethyl glucuronide, ethyl sulphate and fatty acid ethyl esters) after experimental administration of increasing doses of alcohol in adult subjects.

Subjects will be genotyped for genetic polymorphisms of proteins related to ethanol metabolism and effects (as alcohol dehydrogenase and aldehyde dehydrogenase), and the genotypes will be used to evaluate their influence in the results.

ELIGIBILITY:
Inclusion Criteria:

* Understand and accept the study's procedures and sign an informed consent form
* No evidence of somatic or psychiatric disorders as per past medical history and physical examination
* EKG, blood and urine tests taken before entry into the study within the normal range. Minor and transient abnormalities may be acceptable if, according to the Principal Investigator's criterion and the state of the art, they are felt to have no clinical relevance, entail no danger to the participant, and don't interfere with the product's assessment. These abnormalities and their non-relevance must be specifically justified in writing)
* Body mass index (BMI=weight/heigth2) between 19 and 29 kg/m2, weight between 50 and 100 kg (for the 60 and 80 g doses, subjects will be required to weigh a minimum of 67 kg)
* For premenopausal females, a regular menstrual cycle of 26-32 days duration.
* Social or recreational alcohol consumption of at least 1 unit per day (or its equivalent [7 units] over the whole week) and having experienced drunkenness several times

Exclusion Criteria:

* Evidence of a preexisting condition (including gastrointestinal, liver, or kidney disorders) that may alter the absorption, distribution, metabolism or excretion of the drug or symptoms suggestive of drug-induced gastrointestinal irritation
* Previous psychiatric disorders, alcoholism, abuse of prescription drugs or illegal substances or regular consumption of psychoactive drugs
* Having donated blood or having participated in this same study in the preceding 8 weeks, or having participated in any clinical trial with drugs in the preceding 12 weeks
* Having had any somatic disease or having undergone major surgery in the 3 months prior to inclusion in the trial
* Individuals intolerant or having experienced a severe adverse reaction to alcohol
* Having regularly taken medication in the month before the trial, except for vitamins, herb-based remedies, dietary supplements that if, according to the Principal Investigator or his appointed collaborators' opinion, they pose no threat to the subjects and they won't interfere with the study's objectives. Single doses of symptomatic drugs taken during the week before the experimental session will not constitute an exclusion criterion if it can be assumed that it has been completely eliminated on the day of the experimental session
* Smokers of >10 cigarettes/day
* Consumption of >20 g/day of alcohol (females) or of >40 g/day (males)
* Daily consumption of more than 5 coffees, teas, cola drinks or other stimulant or xanthine-containing beverages in the 3 months prior to inclusion in the study
* Hepatitis B, hepatitis C or human immunodeficiency virus-positive individuals
* Pregnant or lactating women, or those using hormonal or unreliable contraceptive methods during the study period. Complete abstinence, intrauterine devices, double barrier methods or a vasectomized sexual partner will be considered acceptable
* Women with amenorrhea or suffering severe premenstrual syndrome
* Individuals of Asian ascent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2014-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC 0-24h) | From baseline to 24 hours after administration
  Calculation of the AUC for plasma fatty acid ethyl esters (palmitic, stearic, linoleic and oleic acid ethyl esters) concentrations. Blood samples will be obtained baseline and at 0,25, 0,50, 0,75,1, 1,25, 1,50, 1,75, 2, 2,5, 3, 3,5, 4, 5, 6, 8, 10, 24h. Additional samples will be collect at 72 h and 1 week, 1 and 2 months after administration. At 3 months a sample will be obtained in selected participants.

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC 0-24h) | From baseline to 24 hours after administration
  Calculation of the AUC for plasma and saliva concentrations of ethanol and its non-oxidative metabolites ethyl sulphate and ethyl glucoronide. Blood samples will be obtained baseline and at 0,25, 0,50, 0,75,1, 1,25, 1,50, 1,75, 2, 2,5, 3, 3,5, 4, 5, 6, 8, 10, 24. Additional samples will be collected at 72 h and 1 week, 1 month and 2 months after administration. At 3 months a sample in selected participants. Saliva samples at baseline and 0,5, 1, 2, 3, 4, 6, 10 and 24 h after administration
Cumulative amount of drug excreted into urine up to collection time of last measurable concentration | From baseline to 72 hours after administration
  Urine will be collected in the following intervals 0-6h, 6-12h, 12-24h, 24-48h, 48-72h and the total amount of ethanol and its non-oxidative metabolites ethyl sulphate and ethyl glucoronide will be calculated.
Elimination half-life | From baseline to 24 hours after administration
  Calculation of elimination half-life from ethanol and its non-oxidative metabolites (fatty acid ethyl esters, ethyl sulphate and ethyl glucoronide) concentrations in plasma
Fatty acid ethyl esters and ethyl glucoronide hair concentrations | Baseline, 1 and 2 months after administration
  Concentrations of fatty acid ethyl esters and ethyl glucoronide in hair at baseline, one and two month after administration. An additional sample at 3 months in selected participants.
Change in subjective effects of ethanol | From baseline to 10 hours after administration
  Participants will self-report their experience on a visual analogue scale of drunkenness and Biphasic alcohol effects scale (BAES) at baseline and 0.5,0.75,1,1.5,2,4,6,8,10 after administration.
Number of Participants with Serious and Non-Serious Adverse Events | From baseline to 24 hours after administration
  Collection of adverse effects spontaneously reported by the participants and/or observed by the investigators
Change in Addiction Research Center Inventory (ARCI) | From baseline to 10 h after administration
  ARCI will be administered baseline and 10 h after administration (subjects should answer at 10 h remembering their experience at the moment of maximum effects)
Change in Evaluation of Subjective Effects of Substances with Abuse Potential (VESSPA) | From baseline to 10 h after administration
  VESSPA will be administered baseline and 10 h after administration (subjects should answer at 10 h remembering their experience at the moment of maximum effects)
Ethanol dose identification questionaire | 10 h after administration
  Participants should guess the dose they have ingested during the experimental session among 5 options (10, 20, 40, 60 and 80 g of ethanol)
Urinary drug concentrations | From 1 week to 2 months
  Urinary concentrations of ethanol and its non-oxidative metabolites ethyl sulphate and ethyl glucoronide will measured at 1 week, 1 and 2 months after administration (3 months in selected subjects)

CONTACTS AND LOCATIONS:
Overall Officials: Francina Fonseca, MD, PhD, Study Director — Parc de Salut Mar; Clara Pérez, MD, PhD, Principal Investigator — Parc de Salut Mar
Locations (1):
- Parc de Salut Mar (IMIM), Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Blaha M, Aaslid R, Douville CM, Correra R, Newell DW. Cerebral blood flow and dynamic cerebral autoregulation during ethanol intoxication and hypercapnia. J Clin Neurosci. 2003 Mar;10(2):195-8. doi: 10.1016/s0967-5868(02)00126-1. PMID 12637048
- [Background] Best CA, Sarkola T, Eriksson CJ, Cluette-Brown JE, Laposata M. Increased plasma fatty acid ethyl ester levels following inhibition of oxidative metabolism of ethanol by 4-methylpyrazole treatment in human subjects. Alcohol Clin Exp Res. 2006 Jul;30(7):1126-31. doi: 10.1111/j.1530-0277.2006.00138.x. PMID 16792559
- [Background] Bottcher M, Beck O, Helander A. Evaluation of a new immunoassay for urinary ethyl glucuronide testing. Alcohol Alcohol. 2008 Jan-Feb;43(1):46-8. doi: 10.1093/alcalc/agm153. Epub 2007 Oct 17. PMID 17942435
- [Background] Cami J, de la Torre R, Garcia-Sevilla L, Ugena B, Knobel H, Segura J. Alcohol antagonism of hypercortisolism induced by naloxone. Clin Pharmacol Ther. 1988 Jun;43(6):599-604. doi: 10.1038/clpt.1988.82. PMID 3378381
- [Background] Di Castelnuovo A, Costanzo S, Bagnardi V, Donati MB, Iacoviello L, de Gaetano G. Alcohol dosing and total mortality in men and women: an updated meta-analysis of 34 prospective studies. Arch Intern Med. 2006 Dec 11-25;166(22):2437-45. doi: 10.1001/archinte.166.22.2437. PMID 17159008
- [Background] Doyle KM, Cluette-Brown JE, Dube DM, Bernhardt TG, Morse CR, Laposata M. Fatty acid ethyl esters in the blood as markers for ethanol intake. JAMA. 1996 Oct 9;276(14):1152-6. PMID 8827968
- [Background] Farre M, de la Torre R, Llorente M, Lamas X, Ugena B, Segura J, Cami J. Alcohol and cocaine interactions in humans. J Pharmacol Exp Ther. 1993 Sep;266(3):1364-73. PMID 8371143
- [Background] Halter CC, Dresen S, Auwaerter V, Wurst FM, Weinmann W. Kinetics in serum and urinary excretion of ethyl sulfate and ethyl glucuronide after medium dose ethanol intake. Int J Legal Med. 2008 Mar;122(2):123-8. doi: 10.1007/s00414-007-0180-8. Epub 2007 Jun 9. PMID 17558515
- [Background] Hoiseth G, Bernard JP, Karinen R, Johnsen L, Helander A, Christophersen AS, Morland J. A pharmacokinetic study of ethyl glucuronide in blood and urine: applications to forensic toxicology. Forensic Sci Int. 2007 Oct 25;172(2-3):119-24. doi: 10.1016/j.forsciint.2007.01.005. Epub 2007 Feb 16. PMID 17306943
- [Background] Hoiseth G, Bernard JP, Stephanson N, Normann PT, Christophersen AS, Morland J, Helander A. Comparison between the urinary alcohol markers EtG, EtS, and GTOL/5-HIAA in a controlled drinking experiment. Alcohol Alcohol. 2008 Mar-Apr;43(2):187-91. doi: 10.1093/alcalc/agm175. Epub 2008 Jan 29. PMID 18230699
- [Background] Holford NH. Clinical pharmacokinetics of ethanol. Clin Pharmacokinet. 1987 Nov;13(5):273-92. doi: 10.2165/00003088-198713050-00001. PMID 3319346
- [Background] Johnson RD, Horowitz M, Maddox AF, Wishart JM, Shearman DJ. Cigarette smoking and rate of gastric emptying: effect on alcohol absorption. BMJ. 1991 Jan 5;302(6767):20-3. doi: 10.1136/bmj.302.6767.20. PMID 1991182
- [Background] Jones MK, Jones BM. Ethanol metabolism in women taking oral contraceptives. Alcohol Clin Exp Res. 1984 Jan-Feb;8(1):24-8. doi: 10.1111/j.1530-0277.1984.tb05026.x. PMID 6370017
- [Background] Kalant H, LeBlanc AE, Wilson A, Homatidis S. Sensorimotor and physiological effects of various alcoholic beverages. Can Med Assoc J. 1975 Apr 19;112(8):953-8. PMID 1131767
- [Background] King AR, Hunter PJ. Alcohol elimination at low blood concentrations among women taking combined oral contraceptives. J Stud Alcohol. 2005 Nov;66(6):738-44. doi: 10.15288/jsa.2005.66.738. PMID 16459935
- [Background] Kopun M, Propping P. The kinetics of ethanol absorption and elimination in twins and supplementary repetitive experiments in singleton subjects. Eur J Clin Pharmacol. 1977;11(5):337-44. doi: 10.1007/BF00566530. PMID 560303
- [Background] Kulig CC, Beresford TP, Everson GT. Rapid, accurate, and sensitive fatty acid ethyl ester determination by gas chromatography-mass spectrometry. J Lab Clin Med. 2006 Mar;147(3):133-8. doi: 10.1016/j.lab.2005.11.006. PMID 16503243
- [Background] Logue PE, Linnoila M, Wallman L, Erwin CW. Effects of ethanol and psychomotor tests on state anxiety: interaction with menstrual cycle in women. Percept Mot Skills. 1981 Apr;52(2):643-8. doi: 10.2466/pms.1981.52.2.643. PMID 7255074
- [Background] Martin E, Moll W, Schmid P, Dettli L. The pharmacokinetics of alcohol in human breath, venous and arterial blood after oral ingestion. Eur J Clin Pharmacol. 1984;26(5):619-26. doi: 10.1007/BF00543496. PMID 6468479
- [Background] Morini L, Marchei E, Vagnarelli F, Garcia Algar O, Groppi A, Mastrobattista L, Pichini S. Ethyl glucuronide and ethyl sulfate in meconium and hair-potential biomarkers of intrauterine exposure to ethanol. Forensic Sci Int. 2010 Mar 20;196(1-3):74-7. doi: 10.1016/j.forsciint.2009.12.035. Epub 2010 Jan 8. PMID 20060246
- [Background] Morfin JP, Kulig C, Everson G, Beresford T. Controlling for serum albumin level improves the correlation between serum fatty acid ethyl esters and blood ethanol level. Alcohol Clin Exp Res. 2007 Feb;31(2):265-8. doi: 10.1111/j.1530-0277.2006.00302.x. PMID 17250618
- [Background] Mumenthaler MS, Taylor JL, O'Hara R, Yesavage JA. Gender differences in moderate drinking effects. Alcohol Res Health. 1999;23(1):55-64. PMID 10890798
- [Background] Nuotto E, Mattila MJ, Seppala T, Konno K. Coffee and caffeine and alcohol effects on psychomotor function. Clin Pharmacol Ther. 1982 Jan;31(1):68-76. doi: 10.1038/clpt.1982.11. PMID 7053307
- [Background] Pragst F, Rothe M, Moench B, Hastedt M, Herre S, Simmert D. Combined use of fatty acid ethyl esters and ethyl glucuronide in hair for diagnosis of alcohol abuse: interpretation and advantages. Forensic Sci Int. 2010 Mar 20;196(1-3):101-10. doi: 10.1016/j.forsciint.2009.12.028. Epub 2010 Jan 12. PMID 20061103
- [Background] Rangno RE, Kreeft JH, Sitar DS. Ethanol 'dose-dependent' elimination: Michaelis-Menten v classical kinetic analysis. Br J Clin Pharmacol. 1981 Nov;12(5):667-73. doi: 10.1111/j.1365-2125.1981.tb01287.x. PMID 7332732
- [Background] Sarkola T, Iles MR, Kohlenberg-Mueller K, Eriksson CJ. Ethanol, acetaldehyde, acetate, and lactate levels after alcohol intake in white men and women: effect of 4-methylpyrazole. Alcohol Clin Exp Res. 2002 Feb;26(2):239-45. PMID 11964564
- [Background] Schroder H, de la Torre R, Estruch R, Corella D, Martinez-Gonzalez MA, Salas-Salvado J, Ros E, Aros F, Flores G, Civit E, Farre M, Fiol M, Vila J, Fernandez-Crehuet J, Ruiz-Gutierrez V, Lapetra J, Saez G, Covas MI; PREDIMED Study Investigators. Alcohol consumption is associated with high concentrations of urinary hydroxytyrosol. Am J Clin Nutr. 2009 Nov;90(5):1329-35. doi: 10.3945/ajcn.2009.27718. Epub 2009 Sep 16. PMID 19759165
- [Background] Soderberg BL, Sicinska ET, Blodget E, Cluette-Brown JE, Suter PM, Schuppisser T, Vetter W, Laposata M. Preanalytical variables affecting the quantification of fatty acid ethyl esters in plasma and serum samples. Clin Chem. 1999 Dec;45(12):2183-90. PMID 10585351
- [Background] Wurst FM, Skipper GE, Weinmann W. Ethyl glucuronide--the direct ethanol metabolite on the threshold from science to routine use. Addiction. 2003 Dec;98 Suppl 2:51-61. doi: 10.1046/j.1359-6357.2003.00588.x. PMID 14984242
- [Background] Wurst FM, Wiesbeck GA, Metzger JW, Weinmann W. On sensitivity, specificity, and the influence of various parameters on ethyl glucuronide levels in urine--results from the WHO/ISBRA study. Alcohol Clin Exp Res. 2004 Aug;28(8):1220-8. doi: 10.1097/01.alc.0000134230.21414.11. PMID 15318121